CLINICAL TRIAL: NCT01322581
Title: A Longitudinal Systems Biological Analysis of Naturally Acquired Malaria Immunity in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911126; 11-I-N126
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Malaria
Keywords: Plasmodium; PBMC; Natural History; Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- observational cohort: This observational-cohort study of individuals (3 months and 40 years of age) will be conducted in the rural village of Kalifabougou, Mali, where Pf transmission is intense and seasonal

SUMMARY:
Plasmodium falciparum (Pf) malaria remains a major cause of morbidity and mortality worldwide. A malaria vaccine would contribute towards efforts to control and eliminate malaria. Optimism that an effective malaria vaccine can be developed is derived in part from the observation that repeated Pf infections can induce protective immunity; however, the mechanisms underlying acquired malaria immunity remain unclear. The goal of the current study is to apply systems biological tools to an observational cohort in an area of intense seasonal Pf transmission to gain insight into the mechanisms underlying naturally acquired malaria immunity. This year-long observational-cohort study of 700 individuals (3 months and 25 years of age) will be conducted in the rural village of Kalifabougou, Mali, where Pf transmission is intense and seasonal. Asymptomatic Pf infection and malaria episodes will be detected by passive and active surveillance. Immune parameters of malaria-protected and -susceptible individuals will be assayed from blood samples collected at strategic time points relative to the malaria season. The primary objective is to identify genome-wide expression profiles induced by Pf infection that are associated with protection from malaria. Secondary objectives include identifying age-related (surrogate for cumulative Pf exposure) changes in Pf-induced gene-expression and serum cytokine profiles, and examining Pf-specific antibody profiles that are associated with protection from malaria using a protein microarray representing 2000 Pf proteins (40 percent of the Pf proteome). Exploratory objectives for this study are to compare the magnitude and quality of the Pf-specific CD4 plus T cell response in malaria-protected and -susceptible individuals and determine how this response varies with age and among individuals before, during, and after malaria season, as well as compare various immune parameters in Pf-infected and uninfected individuals at the end of the dry season to investigate host immune factors associated with chronic asymptomatic Pf infection....

DETAILED DESCRIPTION:
Plasmodium falciparum (Pf) malaria remains a major cause of morbidity and mortality worldwide. A malaria vaccine would contribute towards efforts to control and eliminate malaria. Optimism that an effective malaria vaccine can be developed is derived in part from the observation that repeated Pf infections can induce protective immunity; however, the mechanisms underlying acquired malaria immunity remain unclear. The goal of the current study is to apply systems biological tools to an observational cohort in an area of intense seasonal Pf transmission to gain insight into the mechanisms underlying naturally acquired malaria immunity. This observational-cohort study of individuals (3 months and 40 years of age) will be conducted in the rural village of Kalifabougou, Mali, where Pf transmission is intense and seasonal. Asymptomatic Pf infection and malaria episodes will be detected by passive and active surveillance. Immune parameters of malaria-protected and -susceptible individuals will be assayed from blood samples collected at strategic time points relative to the malaria season. The primary objective is to identify genome-wide expression profiles induced by Pf infection that are associated with protection from malaria. Secondary objectives include identifying age-related (surrogate for cumulative Pf exposure) changes in Pf-induced gene-expression and serum cytokine profiles, and examining Pf-specific antibody profiles that are associated with protection from malaria using a protein microarray representing 2000 Pf proteins (approximately 40% of the Pf proteome). Exploratory objectives for this study are to compare the magnitude and quality of the Pf-specific CD4+ T cell response in malaria-protected and -susceptible individuals and determine how this response varies with age and among individuals before, during, and after malaria season, as well as compare various immune parameters in Pf-infected and uninfected individuals at the end of the dry season to investigate host immune factors associated with chronic asymptomatic Pf infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals 3 months to 40 years of age are eligible to enter the study if they agree to:

* Live in Kalifabougou for the duration of the study (12 months).
* Have blood specimens stored for future studies.

EXCLUSION CRITERIA:

The following eligibility criteria are exclusionary:

* Anemia (hemoglobin less than 7 g/dL).
* Current use of antimalarials, corticosteroids, or other immuno-suppressants.
* Underlying heart disease, bleeding disorder, or other conditions that, in the judgment of the clinical investigators, could increase the risk to the study subjects.
* Fever greater than or equal to 37.5 degrees Celsius or evidence of an acute infection.
* Currently pregnant or planning to become pregnant during the study period.

(Asymptomatic Pf infection at enrollment is not exclusionary).

Ages: 3 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All study subjects will be selected from the village of Kalifabougou, Mali. Male and female volunteers 3 months to 40 years of age will be included. This age range captures the period over which immunity to malaria is acquired in areas of intense Pf transmission like Mali. There is no exclusion based on race, ethnicity, or gender.@@@
Sampling Method: Probability Sample
Enrollment: 1188 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Pf expression profiles | Triannual cross-sectional surveys and convalescence visits
  Identify genome-wide progression profiles induced by Plasmonium falciparum infection that are assocaited with malaria immunity

SECONDARY OUTCOMES:
serum cytokine profiles | Triannual cross-sectional surveys and convalescence visits
  Examine the relationship between age (surrogate for cumulative Pf exposure) and the gene-expression and serum cytokine profilesinduced by Pf infection.
Pf-specific antibody profiles | Triannual cross-sectional surveys and convalescence visits
  Identify Pf-specific antibody profiles that are associated with malaria immunity by using a protein microarray representing 2000 Pf proteins (approx. 40% of the Pf proteome), and determine how these profiles change with age. The objective is to validate and extend findings from a preliminary study performed in the nearby village of Kambila, Mali, where a protein microarray containing approx. 23% of the Pf proteome was used to profile Pf-specific antibody responses in children and adults before and after the 6-month malaria season

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Crompton, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Bamako, Faculty of Medicine, Pharmacy and Odontostomatology, Bamako, Mali

REFERENCES:
- [Background] Tran TM, Aghili A, Li S, Ongoiba A, Kayentao K, Doumbo S, Traore B, Crompton PD. A nested real-time PCR assay for the quantification of Plasmodium falciparum DNA extracted from dried blood spots. Malar J. 2014 Oct 4;13:393. doi: 10.1186/1475-2875-13-393. PMID 25282516
- [Background] Tran TM, Ongoiba A, Coursen J, Crosnier C, Diouf A, Huang CY, Li S, Doumbo S, Doumtabe D, Kone Y, Bathily A, Dia S, Niangaly M, Dara C, Sangala J, Miller LH, Doumbo OK, Kayentao K, Long CA, Miura K, Wright GJ, Traore B, Crompton PD. Naturally acquired antibodies specific for Plasmodium falciparum reticulocyte-binding protein homologue 5 inhibit parasite growth and predict protection from malaria. J Infect Dis. 2014 Mar 1;209(5):789-98. doi: 10.1093/infdis/jit553. Epub 2013 Oct 16. PMID 24133188
- [Background] Doumbo S, Tran TM, Sangala J, Li S, Doumtabe D, Kone Y, Traore A, Bathily A, Sogoba N, Coulibaly ME, Huang CY, Ongoiba A, Kayentao K, Diallo M, Dramane Z, Nutman TB, Crompton PD, Doumbo O, Traore B. Co-infection of long-term carriers of Plasmodium falciparum with Schistosoma haematobium enhances protection from febrile malaria: a prospective cohort study in Mali. PLoS Negl Trop Dis. 2014 Sep 11;8(9):e3154. doi: 10.1371/journal.pntd.0003154. eCollection 2014 Sep. PMID 25210876
- [Derived] Molina-Cruz A, Raytselis N, Withers R, Dwivedi A, Crompton PD, Traore B, Carpi G, Silva JC, Barillas-Mury C. A genotyping assay to determine geographic origin and transmission potential of Plasmodium falciparum malaria cases. Commun Biol. 2021 Sep 30;4(1):1145. doi: 10.1038/s42003-021-02667-0. PMID 34593959
- [Derived] Guha R, Mathioudaki A, Doumbo S, Doumtabe D, Skinner J, Arora G, Siddiqui S, Li S, Kayentao K, Ongoiba A, Zaugg J, Traore B, Crompton PD. Plasmodium falciparum malaria drives epigenetic reprogramming of human monocytes toward a regulatory phenotype. PLoS Pathog. 2021 Apr 6;17(4):e1009430. doi: 10.1371/journal.ppat.1009430. eCollection 2021 Apr. PMID 33822828
- [Derived] Obeng-Adjei N, Larremore DB, Turner L, Ongoiba A, Li S, Doumbo S, Yazew TB, Kayentao K, Miller LH, Traore B, Pierce SK, Buckee CO, Lavstsen T, Crompton PD, Tran TM. Longitudinal analysis of naturally acquired PfEMP1 CIDR domain variant antibodies identifies associations with malaria protection. JCI Insight. 2020 Jun 18;5(12):e137262. doi: 10.1172/jci.insight.137262. PMID 32427581
- [Derived] Liu EW, Skinner J, Tran TM, Kumar K, Narum DL, Jain A, Ongoiba A, Traore B, Felgner PL, Crompton PD. Protein-Specific Features Associated with Variability in Human Antibody Responses to Plasmodium falciparum Malaria Antigens. Am J Trop Med Hyg. 2018 Jan;98(1):57-66. doi: 10.4269/ajtmh.17-0437. PMID 29141757